CLINICAL TRIAL: NCT03265613
Title: Safety and Efficacy of Expanded Allogeneic Adipose-derived Mesenchymal Stem Cells in Patients With Moderate to Severe Psoriasis
Brief Title: Safety and Efficacy of Expanded Allogeneic AD-MSCs in Patients With Moderate to Severe Psoriasis
Acronym: ADMSP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chuanjian Lu, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2017-01
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Mesenchymal Stromal Cells; Psoriasis; Drug Toxicity; Drug Effect
MeSH Terms: conditions — Psoriasis; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AD-MSCs group (Experimental): AD-MSCs（adipose-derived multipotent mesenchymal stem cells ） intravenous injection at a dose of 0.5 million cells/kg at week 0,week 4，week 8 with a duration for treatment for 12 weeks.
  Interventions: Biological: adipose-derived multipotent mesenchymal stem cells

INTERVENTIONS:
Biological: adipose-derived multipotent mesenchymal stem cells — AD-MSCs(adipose-derived multipotent mesenchymal stem cells) were infused intravenously at a dose of 0.5 million cells/kg.
  Other Names: AD-MSCs

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Adipose-derived Mesenchymal Stem Cells (AD-MSCs) with moderate to severe psoriasis. Any adverse events related to AD-MSCs infusion will be monitored. Safety is assessed using incidence of Adverse Events(AEs) and Serious Adverse Events (SAEs). Efficacy is assessed via the proportion of the improvement of PASI (Psoriasis Area and Severity Index), relapse rate in treatment period, changes in PASI score and BSA, as well as DLQI.

DETAILED DESCRIPTION:
Psoriasis is an immune-mediated, genetic disease manifesting in the skin or joints or both. Numerous topical and systemic therapies are available for the treatment of psoriasis. Treatment modalities are chosen on the basis of disease severity, relevant comorbidities, patient preference. For moderate to severe psoriasis, phototherapy, systemic therapy and biologic immune modifying agents are recommended, but all of them have some drawbacks or limitations. Until now, no curative treatment is available. Therefore, it is important to find new treatment for psoriasis.

Mesenchymal stem cells (MSCs) are a kind of adult stem cells that can differentiate into bone, cartilage and adipose cells. Adipos-derived Mesenchymal Stem Cells(AD-MSCs) were isolated from fat tissues and were reported to treat moderate to severe psoriasis vulgaris and psoriasis arthritis successfully by case reports. For the mechanism of the disease, involvement of the immune system in psoriasis is now widely accepted. Mesenchymal stem cells (MSCs) are found to have the function of immunomodulation, migration to skin lesions, limitation of autoimmunity. Therefore, investigators supposed that the injection of AD-MSCs could be beneficial for treatment of moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1．moderate to severe psoriasis vulgaris ( PASI > 10 or BSA >10% ) 2．18 to 65 years old 3．written/signed informed consent

Exclusion Criteria:

1. guttate psoriasis, inverse psoriasis or exclusively associated with the face
2. Acute progressive psoriasis, and erythroderma tendency
3. current (or within 1 year) pregnancy or lactation
4. current significant anxiety or depression with the Self-rating Anxiety Scale (SAS) > 50 or the Self-rating Depression Scale (SDS) > 53, or with other psychiatric disorders
5. With history of primary cardiovascular, respiratory, digestive, urinary, endocrinologic and hematologic diseases, which can't be controlled through ordinary treatments. Those who with malignant diseases, infections, electrolyte imbalance, acid-base disturbance. Patients with clinical test results listed below: abnormal serum calcium level ( Ca2+ > 2.9 mmol/L or < 2 mmol/L);AST or ALT 2 times more than normal upper limit; Creatinine and cystatin C more than normal upper limit; Hemoglobin elevates 20g/L more than normal upper limit,or hemoglobin reduction to anemia; Platelet count less than 75.0*10^9/L; White blood cell less than 3.0*10^9/L; Or any other abnormal laboratory test results, assessed by investigators, that are not suitable for this clinical study
6. Patients with malignant tumors, or when they were enrolled with abnormal tumor markers or with other organ dysfunction
7. allergy to anything else ever before;
8. current registration in other clinical trials or participation within a month;
9. topical treatments (i.e. corticosteroids or retinoic acid or Vitamin D analogs ) within 2 weeks; systemic therapy or phototherapy (ultraviolet radiation B,UVB) and psoralen combined with ultraviolet A (PUVA) within 4 weeks; biological therapy within 12 weeks;
10. medical conditions assessed by investigators, that are not suitable for this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-24 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) related to intervention | 12 weeks (plus or minus 3 days) after treatment
  The proportion of the adverse events related to intervention in the treatment group.
Incidence of serious adverse events (SAEs) related to intervention | 12 weeks (plus or minus 3 days) after treatment
  The proportion of the serious adverse events related to intervention in the treatment group.

SECONDARY OUTCOMES:
Improvement rate of PASI(Psoriasis Area and Severity Index) | 12 weeks (plus or minus 3 days) after treatment
  The proportion of the improvement of PASI(Psoriasis Area and Severity Index) from baseline
PASI(Psoriasis Area and Severity Index) | 12 weeks (plus or minus 3 days) after treatment
  The improvement in PASI score from baseline after treatment
PASI-50 | 12 weeks (plus or minus 3 days) after treatment
  The proportion of patients who achieve at least 50% improvement in PASI score from baseline.
PASI-75 | 12 weeks (plus or minus 3 days) after treatment
  The proportion of patients who achieve at least 75% improvement in PASI score from baseline.
Pruritus Scores on the Visual Analogue Scale | 12 weeks (plus or minus 3 days) after treatment
  Pruritus Scores on the Visual Analogue Scale
BSA | 12 weeks (plus or minus 3 days) after treatment
  the Body Surface Area
DLQI（Dermatology Life Quality Index） | 12 weeks (plus or minus 3 days) after treatment
  the Dermatology Life Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjian Lu, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Yao D, Ye S, He Z, Huang Y, Deng J, Wen Z, Chen X, Li H, Han Q, Deng H, Zhao RC, Lu C. Adipose-derived mesenchymal stem cells (AD-MSCs) in the treatment for psoriasis: results of a single-arm pilot trial. Ann Transl Med. 2021 Nov;9(22):1653. doi: 10.21037/atm-21-5028. PMID 34988162